CLINICAL TRIAL: NCT05194111
Title: Treating Heart Dysfunction Related to Cancer Therapy With Sacubitril/Valsartan (Treat HF)
Brief Title: Treating Heart Dysfunction Related to Cancer Therapy With Sacubitril/Valsartan
Acronym: TREAT-HF
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MCC-21-18830; HM20023601 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2022-01-03; First posted 2022-01-18 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; Heart Dysfunction
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Cardiac magnetic resonance studies will be de-identified and assigned a study number. The identification key will not be available to cardiac magnetic resonance readers so that they are blinded to treatment allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Sacubitril-valsartan (Experimental): Sacubitril-valsartan administered orally twice daily at a maximally tolerate dose (max dose 97mg/103mg twice daily).
  Interventions: Drug: Sacubitril-valsartan
- Arm 2: Valsartan (Experimental): Valsartan administered orally twice daily at a maximally tolerate dose (max dose 160mg twice daily)
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Sacubitril-valsartan — Administered orally twice daily at a maximally tolerate dose (max dose 97mg/103mg twice daily).
  Arms: Arm 1: Sacubitril-valsartan
Drug: Valsartan — Administered orally twice daily at a maximally tolerate dose (max dose 160mg twice daily)
  Arms: Arm 2: Valsartan

SUMMARY:
To determine feasibility of recruitment and tolerability of treatment with sacubitril-valsartan among adult age survivors of cancer diagnosed at or before age 39 who have stage B heart failure.

DETAILED DESCRIPTION:
The current study will test the hypothesis that among adult age survivors of cancer diagnosed at age < 39 years treatment of Stage B heart failure with sacubitril-valsartan is feasible and safe.

ELIGIBILITY:
Inclusion Criteria:

* Age </= 39 years old at time of cancer diagnosis
* Clinical records adequate to determine diagnosis and treatment regimen
* Previous anthracycline chemotherapy
* Global longitudinal strain <18% and/or
* L VEF below the institutional lower limit of normal but >/=40% on echocardiogram or cardiac MRI
* No symptoms of heart failure (shortness of breath, fatigue, swelling). Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea (shortness of breath).

Exclusion Criteria:

* -Age <18 years
* Inability to obtain consent from patient or legally authorized representative
* Active acute or chronic psychiatric illness that in the opinion of the investigator may prevent compliance with study instructions
* Limited English or Spanish proficiency that in the opinion of the investigator may prevent understanding the content of the informed consent form or safely completing the study procedures
* Participation in another concurrent intervention study within 30 days or treatment with an investigational drug within 5 half-lives prior to randomization
* Greater than mild mitral or aortic valve regurgitation/stenosis known pre-cancer therapy
* Severe kidney disease (GFR <30 mL/min/1.73m2)
* Chronic hyperkalemia (>5mmol/L)
* Evidence of COVID-19 within the last 60 days or recent (21 days) exposure to close personal contact with COVID-19.
* Greater than moderate tricuspid or pulmonary valve regurgitation/stenosis known pre-cancer therapy
* Hemodynamically significant congenital heart disease in the opinion of the investigator (not including PFO/small ASD or small VSD)
* Greater than moderate pericardial effusion
* Constrictive cardiomyopathy diagnosed pre-cancer therapy
* Family history of genetic cardiomyopathy
* Evidence of infiltrative cardiomyopathy
* Symptomatic heart disease based on NYHA classification
* Allergy to valsartan or sacubitril
* Inability to complete CMR or 6-minute walk test
* Inability to measure non-invasive blood pressure and heart rate in the ambulatory/home setting
* Pregnant/lactating
* History of severe hypersensitivity reactions to gadolinium-based contrast agents (will perform limited cardiac imaging without contrast)
* Concomitant use of other ACE inhibitors or ARBs, aliskiren, NSAIDs or lithium or the inability to stop these medications for the study

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Determine feasibility of recruitment to this pilot trial by evaluating the eligibility requirements among adult age survivors of cancer diagnosed at or before age 39 who have stage B heart failure. | 24 Months
  Number of participants screened for the clinical trial.
Determine the feasibility of recruitment to this pilot trial by evaluating the eligibility requirements among adult age survivors of cancer diagnosed at or before age 39 who have stage B heart failure. | 27 Months
  Number of participants enrolled on the trial
Determine tolerability of treatment with sacubitril-valsartan among adult age survivors of cancer diagnosed at or before age 39 who have stage B heart failure. | 27 Months
  Number of participants that complete therapy

SECONDARY OUTCOMES:
Evaluate early efficacy of sacubitril-valsartan in the treatment of stage B heart failure among survivors of cancer diagnosed at or before age 39. | 27 Months
  Number of deaths while on study due to cardiac event
Evaluate early efficacy of sacubitril-valsartan in the treatment of stage B heart failure among survivors of cancer diagnosed at or before age 39. | 90 Days
  Number of deaths while on study due to non-cardiac events
Evaluate early efficacy of sacubitril-valsartan in the treatment of stage B heart failure among survivors of cancer diagnosed at or before age 39. | 30 Days
  By the number of Adverse events at 30 days
Evaluate early efficacy of sacubitril-valsartan in the treatment of stage B heart failure among survivors of cancer diagnosed at or before age 39. | 60 Days
  By the number of Adverse events at 60 days
Evaluate early efficacy of sacubitril-valsartan in the treatment of stage B heart failure among survivors of cancer diagnosed at or before age 39. | 90 Days
  By the number of Adverse events at 90 days
Evaluate early efficacy of sacubitril-valsartan in the treatment of stage B heart failure among survivors of cancer diagnosed at or before age 39. | 90 Days
  By determining number of participants with interval change utilizing a 6-minute walk test distance
Evaluate early efficacy of sacubitril-valsartan in the treatment of stage B heart failure among survivors of cancer diagnosed at or before age 39. | 90 Days
  By number of participants with cardiovascular magnetic resonance imaging assessment change in cardiac fibrosis burden.
Evaluate early efficacy of sacubitril-valsartan in the treatment of stage B heart failure among survivors of cancer diagnosed at or before age 39. | 90 Days
  By number of participants with cardiovascular magnetic resonance imaging assessment change in microvascular perfusion.
Evaluate early efficacy of sacubitril-valsartan in the treatment of stage B heart failure among survivors of cancer diagnosed at or before age 39. | 90 Days
  By number of participants with cardiovascular magnetic resonance imaging assessment change in arterial stiffness/4D flow.
Evaluate early efficacy of sacubitril-valsartan in the treatment of stage B heart failure among survivors of cancer diagnosed at or before age 39. | 90 Days
  By number of participants with cardiovascular magnetic resonance imaging assessment change in left ventricular ejection fraction.
Evaluate early efficacy of sacubitril-valsartan in the treatment of stage B heart failure among survivors of cancer diagnosed at or before age 39. | 90 Days
  By number of participants with cardiovascular magnetic resonance imaging assessment change in change in left ventricular strain.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Bottinor, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to make individual participant data available to other researchers at this time.